CLINICAL TRIAL: NCT05943366
Title: Exploring the Feasibility of a Digital Service to Improve Nutrition and Hydration Status of Older Adults: a Mixed-methods Study
Brief Title: Exploring the Feasibility of a Digital Service to Improve Nutrition and Hydration Status of Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chloe French (Other)
Responsible Party: Sponsor-Investigator, Chloe French, Principal Investigator, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17372
Record Dates: First submitted 2023-05-31; First posted 2023-07-13 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Malnutrition; Healthy Aging; Dehydration
Keywords: feasibility; malnutrition; dehydration; digital health
MeSH Terms: conditions — Malnutrition; Dehydration

STUDY DESIGN:
Intervention Model Description: Prior to completing baseline measures, participants will be randomised in a 1:1 ratio to receive the intervention (KOKU-Nut) or to the control group and receive usual care. Randomisation will be undertaken by a separate member of the research team using the Sealed Envelope randomisation service.
Masking Description: Given the nature of the intervention, participants and researchers will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KOKU-Nut (Experimental): Participants will be helped to download KOKU-Nut onto their ipad or tablet during the baseline visit and will receive training. In cases where participants do not have the necessary devices or data to join the intervention, a tablet with KOKU-Nut installed will be provided for the duration of the intervention. Participants will be asked to engage with KOKU-Nut at least 3 times a week throughout the 12-week period.
  Interventions: Device: Keep-on-Keep-Up Nutrition (KOKU-Nut)
- Usual care (No Intervention): Participants will continue with usual care and will receive a leaflet developed by Age UK about the importance of a healthy lifestyle including information on the importance of staying active and nutrition.

INTERVENTIONS:
Device: Keep-on-Keep-Up Nutrition (KOKU-Nut) — Keep-on-Keep-Up (KOKU) is a free, tablet-based strength and balance exercise application that was soft launched in 2020 (https://kokuhealth.com/). KOKU is approved by the National Health Service (NHS) and Organisation for the Review of Care and Health Apps (ORCHA) as a lifestyle app and has been viewed positively by older adults after 6 weeks of independent use. KOKU-Nut is the latest development of this interactive platform and includes nutritional games based on the UK dietary guidelines to nudge older adults to improve their diet with a specific focus on protein, fibre and fluid.
  Arms: KOKU-Nut

SUMMARY:
Trial Design: This is a feasibility randomised controlled trial.

Aim: The study aims to assess the feasibility of conducting a randomised controlled trial using a digital health tool (Keep-On-Keep-Up Nutrition, KOKU-Nut) to improve dietary intake in community-dwelling older adults.

Objectives:

1. Is it feasible and practical to run KOKU-Nut study as a powered randomised controlled trial.
2. Adherence to the intervention, motivations, barriers and facilitators of engaging with KOKU-Nut

Study population:

Community-dwelling adults aged 65 and older

Intervention:

Participants in the intervention group will be asked to engage with KOKU-Nut at least 3 times a week throughout the 12-week period. A crib sheet and contact details for the research team will be available if participants require additional support to help with technical issues.

Control:

Participants will continue with usual care and receive a leaflet developed by Age UK about the importance of a healthy lifestyle.

Timing and duration 3 month intervention with interviews carried out approximately one week after the intervention period

DETAILED DESCRIPTION:
Background:

Dietary patterns can play an important role in health in older age. Apps that encourage dietary change are available and commonly used in younger populations, however; few are designed for the nutritional and technical requirements of older adults. Keep-On-Keep-Up Nutrition (KOKU-Nut) is the latest development of the digital tool and includes nutritional games based on the Eatwell guide to nudge older adults to improve their diet with a specific focus on protein, fibre and fluid. The innovation process has brought together researchers, clinicians, software designers and older users to co-develop the digital tool.

In this study, researchers will test the practicality of KOKU-Nut as an intervention before further larger studies are conducted to assess it's effectiveness.

The aim of this study is to assess the feasibility of conducting a randomised controlled trial using this digital health tool (KOKU-Nut) to improve dietary intake in community-dwelling older adults. Participants will be randomised to receive usual care and an information booklet about living a healthy lifestyle or to the intervention group and asked to engage with KOKU-Nut 3 times a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Living independently in the community
* Have access to the internet (to complete online dietary assessment)
* Willing to use an iPad or tablet (their own or one provided) for the duration of the study

Exclusion Criteria:

* Unable to communicate in English
* Have a known cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported use of KOKU | 12 weeks
  Participants asked about their engagement with KOKU as part of the follow up case report. Participants respond with the option that suits their use best from the following options: every day; 3-4 times a week; 1-2 times a week; once or twice a month
Recruitment rates | 6 months
  Cumulative recruitment against target rate each month
Retention rates | 12 weeks
  Calculated as the number of participants who completed the study divided by the number of participants randomised
Acceptability of the intervention and study design | 12-16 weeks
  This will be assessed qualitatively through semi-structured one-to-one interviews with a subset of participants
Acceptability of the intervention | 12 weeks
  A questionnaire developed by the research team along with the 11-item, 7-point modified treatment evaluation inventory. Higher scores indicate higher acceptability, with a score of 44 indicating moderate acceptability
Usability of the intervention | 12 weeks
  Participants in intervention group will complete the 10-item system usability scale (SUS) to assess perceived usability of the intervention. Responses are measured on a 5-point Likert scale ranging from one (strongly disagree) to five (strongly agree). A score >68 is considered above average usability and >80 is considered high usability.

SECONDARY OUTCOMES:
Change in dietary intake | Baseline, 12 weeks
  Intake of food groups will be generated from a 3-day food diary inputted onto Intake24 software to identify adherence to the Eatwell guide.
Risk of malnutrition | Baseline, 12 weeks
  The malnutrition universal screening tool (MUST) will also be used to assess risk of malnutrition based on BMI, unplanned weight loss and acute disease effect. For each component participants receive a score between 0-2 and cumulative scores are calculated (which can range from 0-6) such that 0 indicates low risk, 1 indicates medium risk and a score of 2 or more indicates a high risk of malnutrition.
Risk of malnutrition | Baseline, 12 weeks
  The Global Leadership Initiative on Malnutrition (GLIM) diagnostic criteria will also be used to assess risk of malnutrition. Participants are assessed on 3 phenotypic criteria (non-volitional weight loss, low body mass index, and reduced muscle mass) and 2 etiologic criteria (reduced food intake or assimilation, and inflammation of disease burden). To diagnose malnutrition at least 1 phenotypic criterion and 1 etiologic criterion should be present.
Change in physical function | Baseline, 12 weeks
  Participants will be instructed to rise from a chair 5 times as quickly as possible with arms folded across their chest and the researcher will record the time taken to complete the task. The researcher will then calculate lower limb muscle power using a validated equation.
Change in physical function | Baseline, 12 weeks
  Grip strength (kg) will be assessed on a Jamar hydraulic dynamometer three times on each hand with the best score used for analysis
Change in health related quality of life | Baseline, 12 weeks
  The EuroQol visual analogue scale (EQ-VAS) will be used for participants to describe their perceived state of health. The score can range from 0 (lowest level of health) to 100 (best health imaginable) where participants indicate how they perceive their current health status both on a number line and numerically.
Change in health related quality of life | Baseline, 12 weeks
  The participants perceived state of health and quality of life will be assessed using the validated EuroQol- 5 Dimension (EQ-5D-5L). The EQ-5D-5Lcomprises five questions assessing mobility, self-care, usual activities, pain or discomfort and anxiety or depression to produce an overall score representing the participant's health profile. The score ranges from one (full health) to zero (state of health equitable to death) with the option to have negative values that indicates a state of health considered to be worse than death
Change in BMI | Baseline, 12 weeks
  Body weight [kg] and height [m] to calculate body mass index (BMI)
Participants socio-demographic characteristics | Baseline
  Age, gender, marital status, occupation, education, income, ethnicity, smoking status, use of digital technology, shopping and cooking habits.
Change in mood | Baseline, 12 weeks
  Participants will complete the 4-item Geriatric depression scale as part of the baseline and follow-up questionnaire. A cumulative scores of 0 indicates participant is not depressed, a score of 1 shows uncertainty and a score between 2 and 4 (inclusive) indicates the participant is depressed.
Change in frailty status | Baseline, 12 weeks
  Researcher will assess frailty of participants based on descriptions and images included in the clinical frailty scale. Scores range from 1 (very fit) to 9 (terminally ill) and a score 5 or more indicates frailty.
Adverse events | From recruitment until study end (approximately 14 weeks)
  Number of adverse events that occurred as a result of participation in the study

CONTACTS AND LOCATIONS:
Overall Officials: Emma Stanmore, Principal Investigator — University of Manchester
Locations (1):
- Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] French C, Burden S, Stanmore E. Digital Intervention (Keep-On-Keep-Up Nutrition) to Improve Nutrition in Older Adults: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 30;13:e50922. doi: 10.2196/50922. PMID 38687981